CLINICAL TRIAL: NCT00211705
Title: Management of Elevated Cholesterol in the Primary Prevention Group of Adult Japanese(MEGA Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mitsukoshi Health and Welfare Foundation (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry); Ministry of Health, Labour and Welfare, Japan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEGA
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2005-06

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia; coronary heart disease; prevention; stroke; pravastatin
MeSH Terms: conditions — Hyperlipidemias; Coronary Disease; Stroke | interventions — Diet

INTERVENTIONS:
Behavioral: Diet
Drug: Diet+pravastatin

SUMMARY:
To evaluate the primary preventive effect of low-dose pravastatin against coronary heart disease (CHD) in Japanese hypercholesterolemic patients.

DETAILED DESCRIPTION:
MEGA Study is the first prospective, randomized, controlled trial conducted in Japan to evaluate the primary preventive effect of pravastatin against CHD in daily clinical practice. Because the dose of pravastatin used in the MEGA Study was 10-20 mg/day, which is consistent with the approved doses in Japan and lower than the doses used in previous large-scale clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* TC:220～270mg/dl
* Male: 40-70 years old/ female: postmenopausal-70 years old
* <40kg in weight

Exclusion Criteria:

* FH
* History of CHD(angina, MI, post-PTCA/CABG, etc.)
* History of CVA(stroke, TIA, etc.)
* Underlying malignant tumor

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000
Dates: Start 1994-02; Study Completion 2004-03

PRIMARY OUTCOMES:
Coronary Heart Disease(CHD)[fatal/non-fatal MI, sudden/cardiac death, angina, revascularization]

SECONDARY OUTCOMES:
Stroke, cerebrovascular infarction(CI), CHD+CI, all cardiovascular events, total mortality

CONTACTS AND LOCATIONS:
Overall Officials: Haruo Nakamura, MD, Study Chair — Mitsukoshi Health and Welfare

REFERENCES:
- [Background] Management of Elevated Cholesterol in the Primary Prevention Group of Adult Japanese (MEGA) Study Group. Design and baseline characteristics of a study of primary prevention of coronary events with pravastatin among Japanese with mildly elevated cholesterol levels. Circ J. 2004 Sep;68(9):860-7. doi: 10.1253/circj.68.860. PMID 15329509
- [Result] Nakamura H, Arakawa K, Itakura H, Kitabatake A, Goto Y, Toyota T, Nakaya N, Nishimoto S, Muranaka M, Yamamoto A, Mizuno K, Ohashi Y; MEGA Study Group. Primary prevention of cardiovascular disease with pravastatin in Japan (MEGA Study): a prospective randomised controlled trial. Lancet. 2006 Sep 30;368(9542):1155-63. doi: 10.1016/S0140-6736(06)69472-5. PMID 17011942
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702
- [Derived] Nakamura H, Mizuno K; MEGA Study Group. Cardiovascular and cancer events in hyper-high-density lipoprotein cholesterolemic patients: a post hoc analysis of the MEGA study. Lipids Health Dis. 2014 Aug 18;13:133. doi: 10.1186/1476-511X-13-133. PMID 25135178
- [Derived] Tajima N, Kurata H, Ohashi Y, Mizuno K, Nakamura H. Management of Elevated Cholesterol in the primary prevention Group of Adult Japanese (MEGA) Study assists the view that a fasting plasma glucose level >/=100 mg/dL increases cardiovascular risk. J Diabetes Investig. 2011 Oct 7;2(5):399-405. doi: 10.1111/j.2040-1124.2011.00121.x. PMID 24843520
- [Derived] Matsushima T, Nakaya N, Mizuno K, Ohashi Y, Teramoto T, Yokoyama S, Ichikawa S, Ishikura N, Kamiyama K, Nakamura H; MEGA Study Group. The effect of low-dose pravastatin in metabolic syndrome for primary prevention of cardiovascular disease in Japan: a post hoc analysis of the MEGA study. J Cardiovasc Pharmacol Ther. 2012 Jun;17(2):153-8. doi: 10.1177/1074248411421777. Epub 2011 Oct 3. PMID 22573644
- [Derived] Nakaya N, Mizuno K, Ohashi Y, Teramoto T, Yokoyama S, Hirahara K, Mizutani M, Nakamura H; MEGA Study Group. Low-dose pravastatin and age-related differences in risk factors for cardiovascular disease in hypercholesterolaemic Japanese: analysis of the management of elevated cholesterol in the primary prevention group of adult Japanese (MEGA study). Drugs Aging. 2011 Sep 1;28(9):681-92. doi: 10.2165/11595620-000000000-00000. PMID 21815708
- [Derived] Kushiro T, Mizuno K, Nakaya N, Ohashi Y, Teramoto T, Yokoyama S, Kakinoki S, Nakamura H; MEGA Study Group. Blood pressure control status and effects of pravastatin on cardiovascular events occurrence in patients with dyslipidaemia. J Hum Hypertens. 2012 Jun;26(6):388-95. doi: 10.1038/jhh.2011.49. Epub 2011 May 19. PMID 21593784
- [Derived] Nakamura H, Mizuno K, Ohashi Y, Yoshida T, Hirao K, Uchida Y; MEGA Study Group. Pravastatin and cardiovascular risk in moderate chronic kidney disease. Atherosclerosis. 2009 Oct;206(2):512-7. doi: 10.1016/j.atherosclerosis.2009.03.031. Epub 2009 Apr 5. PMID 19423108
- [Derived] Kushiro T, Mizuno K, Nakaya N, Ohashi Y, Tajima N, Teramoto T, Uchiyama S, Nakamura H; Management of Elevated Cholesterol in the Primary Prevention Group of Adult Japanese Study Group. Pravastatin for cardiovascular event primary prevention in patients with mild-to-moderate hypertension in the Management of Elevated Cholesterol in the Primary Prevention Group of Adult Japanese (MEGA) Study. Hypertension. 2009 Feb;53(2):135-41. doi: 10.1161/HYPERTENSIONAHA.108.120584. Epub 2008 Dec 22. PMID 19104004
- [Derived] Mizuno K, Nakaya N, Ohashi Y, Tajima N, Kushiro T, Teramoto T, Uchiyama S, Nakamura H; MEGA Study Group. Usefulness of pravastatin in primary prevention of cardiovascular events in women: analysis of the Management of Elevated Cholesterol in the Primary Prevention Group of Adult Japanese (MEGA study). Circulation. 2008 Jan 29;117(4):494-502. doi: 10.1161/CIRCULATIONAHA.106.671826. Epub 2008 Jan 2. PMID 18172039